CLINICAL TRIAL: NCT02828969
Title: Clinical Trajectory of Children and Adolescents With Disruptive Behavior Admitted to Pediatric and Psychiatric Emergencies.
Brief Title: Clinical and Social Trajectory of Children and Adolescents With Disruptive Behavior
Acronym: TRAJECTORY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL16_0432
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Disruptive Behavior
Keywords: Trajectory; Emergency room; Conduct disorder; Care management
MeSH Terms: conditions — Problem Behavior; Emergencies; Conduct Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children and adolescents with conduct disorders (Other): Girls and boys having less than 18 years old and admitted to emergency room for aggressiveness, violence, fugue or theft.
  Interventions: Other: Phone call or physical consultation

INTERVENTIONS:
Other: Phone call or physical consultation

SUMMARY:
Conduct disorders are defined as "repetitive and persistent pattern of behavior in which the basic rights of others or major age-appropriate norms are violated". So defined, these disorders are at the crossroads of psychiatry, social field and justice. Conduct disorder management is a public health issue and a societal question. Conduct disorders affect 5 to 9% of 15-year old boys.

Care management of children and adolescents admitted for disruptive behaviors in emergency rooms is an issue. No consensus or official recommendation exists. However, use of emergency care in this context is increasing in most western countries and it exposes to several risks (inappropriate use of hospitalizations, social rupture, ignorance of comorbidities and suicide risk). The Trajectories project is designed to describe children and adolescents with disruptive behaviors, their care management and to follow their life trajectory and psychiatric evolution after admission to emergency rooms. Better understanding this population will improve their medical and social care management, thereby giving professionals the right tools.

The main objective of this project is to implement a multidisciplinary and integrative research combining clinical considerations and social sciences to determine the "trajectory" of this population.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents admitted to emergency rooms for aggressiveness, violence, fugue or theft

Exclusion Criteria:

* Children and adolescents admitted to emergency rooms for a reason not directly link with aggressiveness, violence, fugue or theft
* Opposition to the subject or the family to participate to this research

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Description of the children and adolescents admitted to emergency rooms for aggressiveness, violence, fugue or theft. | At inclusion
  This study is intended to characterized the population of children and adolescents admitted to emergency rooms for disruptive behavior

SECONDARY OUTCOMES:
Nature and type of the care management provided to children and adolescents admitted to emergency rooms for disruptive behavior | At inclusion
  Type of care management (hospitalization, reason of admission, type of caregiver at the admission, perception of the care management…)
description of patients' perceptions of the care management | at inclusion
  the patients' perceptions of the care management will be evaluated by the Score at the rating scale (1 to 10) evaluating perceptions support to emergencies.
description of patients' perceptions of the care management | 6 months
  the patients' perceptions of the care management will be evaluated by the Score at the rating scale (1 to 10) evaluating perceptions support to emergencies.
description of patients' perceptions of the care management | 12 months
  the patients' perceptions of the care management will be evaluated by the Score at the rating scale (1 to 10) evaluating perceptions support to emergencies.
description of patients' perceptions of the care management | 24 months
  the patients' perceptions of the care management will be evaluated by the Score at the rating scale (1 to 10) evaluating perceptions support to emergencies.
Identification of patients'psychiatric underlying disorders | At 6 months
  The patients'psychiatric underlying disorders will be evaluated by Psychiatric diagnosis : criteria of ICD (International Classification of Diseases) 10
Social and clinical evolution after the initial admission to emergency room | 6 months
  The social evolution will be evaluated by social rupture, exclusion, penal measure and the clinical evolution will be evaluated by suicide attempt, disruptive behavior recurrence….
Social and clinical evolution after the initial admission to emergency room | 12 months
  The social evolution will be evaluated by social rupture, exclusion, penal measure and the clinical evolution will be evaluated by suicide attempt, disruptive behavior recurrence….
Social and clinical evolution after the initial admission to emergency room | 24 months
  The social evolution will be evaluated by social rupture, exclusion, penal measure and the clinical evolution will be evaluated by suicide attempt, disruptive behavior recurrence….

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon/bron, France

IPD SHARING:
Plan to Share IPD: No